CLINICAL TRIAL: NCT03638596
Title: Leveraging Transdermal Alcohol Monitoring to Reduce Drinking Among DWI Defendants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20160425H; 5R01AA014988 (NIH)
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Drunk Driving
Keywords: Alcohol Impaired Driving; Driving While Intoxicated; Driving Under the Influence; Driving While Impaired
MeSH Terms: conditions — Driving Under the Influence

STUDY DESIGN:
Intervention Model Description: random assignment to treatment and control arms
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingency Management (Experimental): Incentive delivery contingent upon maintaining transdermal alcohol concentration below cut-off
  Interventions: Behavioral: Contingency Management
- Control (Placebo Comparator): Incentive delivery not contingent on transdermal alcohol concentration
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Contingency Management — Incentive provided for changing alcohol drinking patterns based on ankle monitor
  Arms: Contingency Management
Behavioral: Control — Incentive provided is not contingent on alcohol drinking patterns based on ankle monitor
  Arms: Control

SUMMARY:
The current study will evaluate the efficacy of contingency management (i.e., reinforcement for avoiding heavy drinking) among adults arrested for drunk driving and who are at risk for ongoing heavy drinking.

DETAILED DESCRIPTION:
Individuals who have a drunk driving arrest and are at risk for ongoing heavy drinking will be recruited to test the efficacy of contingency management for reducing alcohol use and identifying mechanisms of change. We will recruit those arrested for drunk driving offenses, ≥ 21 years of age, who at risk for ongoing heavy alcohol use and randomize them to one of two groups: control or a contingency management. Participants experience 8 weekly assessments of current alcohol use and other variables associated with changes in alcohol use. Post-intervention, participants will return to the laboratory once per month at 3, 6, 9, and 12 months post-study entry for follow-up procedures to determine the mechanisms of drinking behavior change.

ELIGIBILITY:
Inclusion Criteria:

* arrested for drunk driving offense

Exclusion Criteria:

* significant alcohol withdrawal symptoms
* medical condition that would contraindicate participation (e.g., pregnancy, scheduled surgery)
* inability to comprehend the informed consent process or study instructions
* presence of a DSM-5 psychiatric disorder with symptoms of psychosis and/or delirium
* incarceration

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Percent heavy drinking days | 8-weeks
  Percent of days with estimated breath alcohol concentration .08% or higher or self-reported drinks > 5 for men and > 4 for women

SECONDARY OUTCOMES:
Percent drinking days | 8-weeks
  Percent of days with any positive transdermal alcohol concentration >.02 or any self-reported drinks
Follow-up percent heavy drinking days | 12-months
  Self-reported drinks > 5 for men and > 4 for women
Follow-up percent drinking days | 12-months
  Any self-reported drinks
Measurement of alcohol biomarker | Baseline to 8-weeks
  Change in phosphatidylethanol (PEth) using an assay on a blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Hill-Kapturczak, PhD, Principal Investigator — The University of Texas Health Science Center San Antonio
Locations (1):
- University of Texas Health Science Center San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No